CLINICAL TRIAL: NCT06368713
Title: Exercise Improves Gastrointestinal Function in Peritoneal Dialysis Patients: A Single Center Prospective Randomized Controlled Study
Brief Title: Exercise Improves Gastrointestinal Function in Peritoneal Dialysis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jin Chen, associate chief physician, Sichuan Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PD-GIEX
Record Dates: First submitted 2024-04-07; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Peritoneal Dialysis; Exercise; Gastrointestinal Function; Quality of Life; Chronic Kidney Diseases
Keywords: Peritoneal Dialysis; Exercise intervention; Gastrointestinal function; Telehealth
MeSH Terms: conditions — Motor Activity; Renal Insufficiency, Chronic | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise intervention group (Experimental): The exercise intervention group will receive guidance for exercises and participate in remote exercise sessions monitored.
  Interventions: Behavioral: Exercise
- Control group (No Intervention): The control group will not receive exercise intervention.

INTERVENTIONS:
Behavioral: Exercise — * Frequency: Exercise sessions will occur no less than three times per week.
  * Intensity: The intensity will be based on a rating of perceived exertion score ranging from 12 to 16 on a scale of 6 to 20.
  * Exercise duration: Each exercise session will last approximately 30 minutes.
  * Exercise Type:The exercise regimen will include aerobic exercise, resistance exercise, and flexibility training.
  Arms: Exercise intervention group

SUMMARY:
This study will investigate the impact of exercise on gastrointestinal function in peritoneal dialysis patients.

DETAILED DESCRIPTION:
Maintaining gastrointestinal health is paramount for individuals on peritoneal dialysis, yet it frequently goes unnoticed within the broader scope of their health management. The effectiveness of dialysis treatments, along with aspects such as nutrient uptake and life quality, can be adversely affected by gastrointestinal disturbances. The volume of fluid within the peritoneal space, medications associated with dialysis, and the procedure of dialysis itself are all known to play roles in modulating gastrointestinal health.

The role of physical activity in enhancing gastrointestinal wellness among those with chronic conditions has gained acknowledgment over time. Customized exercise regimes have been shown to markedly better gastrointestinal symptoms, the efficiency of nutrient absorption, and overall life satisfaction among these patients. Notably, the specific influence of exercise on the gastrointestinal functions of individuals undergoing peritoneal dialysis has yet to be explored.

This investigation aims to assess the effects of exercise on the gastrointestinal health of peritoneal dialysis patients. Participants will be divided equally into an exercise group and a control group, following a randomized selection process. After collecting data throughout a four-month period, an analysis will be conducted to ascertain the benefits of physical activity for enhancing the gastrointestinal function of those on peritoneal dialysis. The outcomes of this study are anticipated to guide clinicians in recommending strategies to improve gastrointestinal health in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have undergone peritoneal dialysis for more than 3 months.
2. Age between 18 and 65 years.
3. Possession of a smartphone and proficiency in its usage.
4. Willingness to provide voluntary informed consent by signing the consent form.

Exclusion Criteria:

1. Recent systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥110 mmHg, or systolic blood pressure ≤90 mmHg or diastolic blood pressure ≤60 mmHg within the past week.
2. Presence of severe cardiovascular diseases, including but not limited to:

   * Heart failure classified as New York Heart Association (NYHA) functional grade IV-V.
   * Severe arrhythmias such as third-degree atrioventricular block, sick sinus syndrome, paroxysmal supraventricular tachycardia, or ventricular tachycardia.
   * Unstable angina.
   * Pulmonary arterial hypertension with pulmonary arterial pressure ≥25 mmHg.
   * Severe pericardial effusion, valve stenosis, hypertrophic cardiomyopathy, or aortic dissection.
3. Severe pulmonary diseases, including but not limited to:

   * Severe chronic obstructive pulmonary disease (COPD).
   * Pulmonary embolism.
   * Lung cancer.
   * Severe pulmonary infection.
4. Presence of deep venous thrombosis.
5. Severe neurological, muscular, bone, or joint diseases that hinder compliance with exercise.
6. Participation in other concurrent exercise programs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in GIQLI | Patients are required to complete the questionnaire at baseline, 2 weeks, 4 weeks, 2 months, and 3 months after the start of the intervention.
  The Gastrointestinal Quality of Life Index is a 36-item questionnaire assessing the impact of gastrointestinal symptoms and diseases on daily life. The GIQLI includes five domains: gastrointestinal symptoms (19 items), emotional status (5 items), physical function (7 items), social function (4 items), and medical inconvenience (1 item). Each item is scored from 0 to 4, with a total score ranging from 0 to 144. Higher scores indicate better quality of life.

SECONDARY OUTCOMES:
Change in GSRS | Patients are also required to complete the questionnaire at baseline, 2 weeks, 4 weeks, 2 months, and 3 months after the start of the intervention.
  Gastrointestinal Symptom Rating Scale (GSRS)consists of 15 questions aimed at assessing the impact of upper and lower gastrointestinal symptoms. It includes five dimensions (symptoms of gastroesophageal reflux, diarrhea, constipation, abdominal pain, and indigestion), with each question scored from 0 (no discomfort) to 6 (very severe discomfort). A GSRS score of ≥1 defines the presence of gastrointestinal symptoms A higher score indicates more severe gastrointestinal symptoms.
Change in PAC-SYM | Patients are required to complete the questionnaire at baseline, 2 weeks, 4 weeks, 2 months, and 3 months after the start of the intervention.
  Patient Assessment of Constipation Symptom (PAC-SYM) comprises 12 questions designed to evaluate the impact of upper and lower gastrointestinal symptoms. It assesses five dimensions, including symptoms of gastroesophageal reflux, diarrhea, constipation, abdominal pain, and indigestion. Each question is scored from 0 (no discomfort) to 6 (very severe discomfort). A GSRS score of ≥1 indicates the presence of gastrointestinal symptoms, with higher scores indicating more severe symptoms.
Change in 6-MWT | Measurements are taken before the start of the intervention, 2 weeks and 3 months after the intervention.
  The 6-Minute Walk Test (6-MWT) is conducted along a 10-meter path marked with two turning points. Patients are instructed to walk back and forth along the path for 6 minutes, and the total walking distance is measured. The test duration is monitored using a stopwatch. Based on the walking distance achieved, patients' heart failure severity is categorized as follows: <150m indicates severe heart failure; 150-425m indicates moderate heart failure; 426-550m indicates mild heart failure.
Change in SGA | Patients are required to complete the SGA scale at the baseline and 3 months after the intervention.
  The Subjective Global Assessment (SGA) is a tool utilized to assess the nutritional status of patients. It involves a comprehensive evaluation of various factors such as weight change, dietary intake, gastrointestinal symptoms, and functional capacity.
Change in measured Gastrointestinal Hormones | Blood samples will be collected at the baseline and and 3 months the intervention.
  The assessment includes the measurement of Ghrelin, Pancreatic polypeptide, and peotideYY, which are gastrointestinal hormones involved in regulating appetite and digestion.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Chen, Doctor, Principal Investigator — Sichuan Academy of Medical Sciences , University of Electronic Science and Technology of China,
Locations (1):
- Sichuan Academy of Medical Sciences and Sichuan Provincial People's Hospital,School of Medicine, University of Electronic Science and Technology of China, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ROB CG, RICHARDSON JS. Peritoneal dialysis. Lancet. 1947 Feb 1;1(6440):195. doi: 10.1016/s0140-6736(47)91172-0. No abstract available. PMID 20341549
- [Background] Zhang P, Wang X, Li S, Cao X, Zou J, Fang Y, Shi Y, Xiang F, Shen B, Li Y, Fang B, Zhang Y, Guo R, Lv Q, Zhang L, Lu Y, Wang Y, Yu J, Xie Y, Wang R, Chen X, Yu J, Zhang Z, He J, Zhan J, Lv W, Nie Y, Cai J, Xu X, Hu J, Zhang Q, Gao T, Jiang X, Tan X, Xue N, Wang Y, Ren Y, Wang L, Zhang H, Ning Y, Chen J, Zhang L, Jin S, Ren F, Ehrlich SD, Zhao L, Ding X. Metagenome-wide analysis uncovers gut microbial signatures and implicates taxon-specific functions in end-stage renal disease. Genome Biol. 2023 Oct 12;24(1):226. doi: 10.1186/s13059-023-03056-y. PMID 37828586
- [Background] Jiang S, Xie S, Lv D, Wang P, He H, Zhang T, Zhou Y, Lin Q, Zhou H, Jiang J, Nie J, Hou F, Chen Y. Alteration of the gut microbiota in Chinese population with chronic kidney disease. Sci Rep. 2017 Jun 6;7(1):2870. doi: 10.1038/s41598-017-02989-2. PMID 28588309
- [Background] Hirako M, Kamiya T, Misu N, Kobayashi Y, Adachi H, Shikano M, Matsuhisa E, Kimura G. Impaired gastric motility and its relationship to gastrointestinal symptoms in patients with chronic renal failure. J Gastroenterol. 2005 Dec;40(12):1116-22. doi: 10.1007/s00535-005-1709-6. PMID 16378175
- [Background] Yi C, Wang X, Ye H, Lin J, Yang X. Patient-reported gastrointestinal symptoms in patients with peritoneal dialysis: the prevalence, influence factors and association with quality of life. BMC Nephrol. 2022 Mar 9;23(1):99. doi: 10.1186/s12882-022-02723-9. PMID 35264119
- [Background] Duncanson E, Chur-Hansen A, Jesudason S. Psychosocial consequences of gastrointestinal symptoms and dietary changes in people receiving automated peritoneal dialysis. J Ren Care. 2019 Mar;45(1):41-50. doi: 10.1111/jorc.12265. Epub 2018 Dec 25. PMID 30585418
- [Background] Strid H, Simren M, Johansson AC, Svedlund J, Samuelsson O, Bjornsson ES. The prevalence of gastrointestinal symptoms in patients with chronic renal failure is increased and associated with impaired psychological general well-being. Nephrol Dial Transplant. 2002 Aug;17(8):1434-9. doi: 10.1093/ndt/17.8.1434. PMID 12147791
- [Background] Setyapranata S, Holt SG. The Gut in Older Patients on Peritoneal Dialysis. Perit Dial Int. 2015 Nov;35(6):650-4. doi: 10.3747/pdi.2014.00341. PMID 26702007
- [Background] Kosmadakis G, Albaret J, da Costa Correia E, Somda F, Aguilera D. Gastrointestinal Disorders in Peritoneal Dialysis Patients. Am J Nephrol. 2018;48(5):319-325. doi: 10.1159/000494145. Epub 2018 Oct 19. PMID 30343294
- [Background] Cha RR, Park SY, Camilleri M; Constipation Research Group of Korean Society of Neurogastroenterology and Motility. Constipation in Patients With Chronic Kidney Disease. J Neurogastroenterol Motil. 2023 Oct 30;29(4):428-435. doi: 10.5056/jnm23133. PMID 37814433
- [Background] Tian N, Li L, Ng JK, Li PK. The Potential Benefits and Controversies of Probiotics Use in Patients at Different Stages of Chronic Kidney Disease. Nutrients. 2022 Sep 29;14(19):4044. doi: 10.3390/nu14194044. PMID 36235699
- [Background] Biruete A, Shin A, Kistler BM, Moe SM. Feeling gutted in chronic kidney disease (CKD): Gastrointestinal disorders and therapies to improve gastrointestinal health in individuals CKD, including those undergoing dialysis. Semin Dial. 2024 Jul-Aug;37(4):334-349. doi: 10.1111/sdi.13030. Epub 2021 Oct 27. PMID 34708456
- [Background] Hamaguchi T, Tayama J, Suzuki M, Nakaya N, Takizawa H, Koizumi K, Amano Y, Kanazawa M, Fukudo S. The effects of locomotor activity on gastrointestinal symptoms of irritable bowel syndrome among younger people: An observational study. PLoS One. 2020 May 29;15(5):e0234089. doi: 10.1371/journal.pone.0234089. eCollection 2020. PMID 32470098
- [Background] Bianco A, Russo F, Franco I, Riezzo G, Donghia R, Curci R, Bonfiglio C, Prospero L, D'Attoma B, Ignazzi A, Campanella A, Osella AR. Enhanced Physical Capacity and Gastrointestinal Symptom Improvement in Southern Italian IBS Patients following Three Months of Moderate Aerobic Exercise. J Clin Med. 2023 Oct 26;12(21):6786. doi: 10.3390/jcm12216786. PMID 37959251
- [Background] Riezzo G, Prospero L, D'Attoma B, Ignazzi A, Bianco A, Franco I, Curci R, Campanella A, Bonfiglio C, Osella AR, Russo F. The Impact of a Twelve-Week Moderate Aerobic Exercise Program on Gastrointestinal Symptom Profile and Psychological Well-Being of Irritable Bowel Syndrome Patients: Preliminary Data from a Southern Italy Cohort. J Clin Med. 2023 Aug 17;12(16):5359. doi: 10.3390/jcm12165359. PMID 37629401
- [Background] Zhang F, Liao J, Zhang W, Wang H, Huang L, Shen Q, Zhang H. Effects of Baduanjin Exercise on Physical Function and Health-Related Quality of Life in Peritoneal Dialysis Patients: A Randomized Trial. Front Med (Lausanne). 2021 Nov 29;8:789521. doi: 10.3389/fmed.2021.789521. eCollection 2021. PMID 34912835
- [Background] Abdelbasset WK, Ibrahim AA, Althomali OW, Hussein HM, Alrawaili SM, Alsubaie SF. Effect of twelve-week concurrent aerobic and resisted exercise training in non-dialysis day on functional capacity and quality of life in chronic kidney disease patients. Eur Rev Med Pharmacol Sci. 2022 Sep;26(17):6098-6106. doi: 10.26355/eurrev_202209_29626. PMID 36111910
- [Background] Weiner DE, Liu CK, Miao S, Fielding R, Katzel LI, Giffuni J, Well A, Seliger SL. Effect of Long-term Exercise Training on Physical Performance and Cardiorespiratory Function in Adults With CKD: A Randomized Controlled Trial. Am J Kidney Dis. 2023 Jan;81(1):59-66. doi: 10.1053/j.ajkd.2022.06.008. Epub 2022 Aug 6. PMID 35944747
- [Background] Deus LA, Correa HL, Neves RVP, Reis AL, Honorato FS, Araujo TB, Souza MK, Haro AS, Silva VL, Barbosa JMDS, Padula IA, Andrade RV, Simoes HG, Prestes J, Stone WJ, Melo GF, Rosa TS. Metabolic and hormonal responses to chronic blood-flow restricted resistance training in chronic kidney disease: a randomized trial. Appl Physiol Nutr Metab. 2022 Feb;47(2):183-194. doi: 10.1139/apnm-2021-0409. Epub 2022 Jan 21. PMID 35062832
- [Background] Li WY, Chiu FC, Zeng JK, Li YW, Huang SH, Yeh HC, Cheng BW, Yang FJ. Mobile Health App With Social Media to Support Self-Management for Patients With Chronic Kidney Disease: Prospective Randomized Controlled Study. J Med Internet Res. 2020 Dec 15;22(12):e19452. doi: 10.2196/19452. PMID 33320101
- [Background] Gravina EPL, Pinheiro BV, da Silva Jesus LA, da Silva LP, da Silva RN, Silva K, de Paula RB, Reboredo MM. Effects of long-term aerobic training and detraining on functional capacity and quality of life in hemodialysis patients: A pilot study. Int J Artif Organs. 2020 Jun;43(6):411-415. doi: 10.1177/0391398819890622. Epub 2019 Nov 27. PMID 31774015
- [Background] Bennett PN, Bohm C, Harasemiw O, Brown L, Gabrys I, Jegatheesan D, Johnson DW, Lambert K, Lightfoot CJ, MacRae J, Meade A, Parker K, Scholes-Robertson N, Stewart K, Tarca B, Verdin N, Wang AY, Warren M, West M, Zimmerman D, Li PK, Thompson S. Physical activity and exercise in peritoneal dialysis: International Society for Peritoneal Dialysis and the Global Renal Exercise Network practice recommendations. Perit Dial Int. 2022 Jan;42(1):8-24. doi: 10.1177/08968608211055290. Epub 2021 Nov 7. PMID 34743628
- [Background] Bennett PN, Bohm C, Yee-Moon Wang A, Kanjanabuch T, Figueiredo AE, Harasemiw O, Brown L, Gabrys I, Jegatheesan D, Lambert K, Lightfoot CJ, MacRae J, Scholes-Robertson N, Stewart K, Tarca B, Verdin N, Warren M, West M, Zimmerman D, Finderup J, Ford E, Ribeiro HS, Xu Q, Thompson S. An International Survey of Peritoneal Dialysis Exercise Practices and Perceptions. Kidney Int Rep. 2023 May 3;8(7):1389-1398. doi: 10.1016/j.ekir.2023.04.024. eCollection 2023 Jul. PMID 37441469
- [Background] Wu HHL, Poulikakos D, Hurst H, Lewis D, Chinnadurai R. Delivering Personalized, Goal-Directed Care to Older Patients Receiving Peritoneal Dialysis. Kidney Dis (Basel). 2023 Jun 23;9(5):358-370. doi: 10.1159/000531367. eCollection 2023 Oct. PMID 37901709
- [Background] Eypasch E, Williams JI, Wood-Dauphinee S, Ure BM, Schmulling C, Neugebauer E, Troidl H. Gastrointestinal Quality of Life Index: development, validation and application of a new instrument. Br J Surg. 1995 Feb;82(2):216-22. doi: 10.1002/bjs.1800820229. PMID 7749697
- [Background] Heine GH, Kastner CY, Jahnke T, Kohler H, Kuhlmann MK. Does a history of peritoneal dialysis result in an impaired gastrointestinal life quality? Hemodial Int. 2007 Oct;11(4):461-7. doi: 10.1111/j.1542-4758.2007.00218.x. PMID 17922745
- [Background] Revicki DA, Wood M, Wiklund I, Crawley J. Reliability and validity of the Gastrointestinal Symptom Rating Scale in patients with gastroesophageal reflux disease. Qual Life Res. 1998 Jan;7(1):75-83. doi: 10.1023/a:1008841022998. PMID 9481153
- [Background] Frank L, Kleinman L, Farup C, Taylor L, Miner P Jr. Psychometric validation of a constipation symptom assessment questionnaire. Scand J Gastroenterol. 1999 Sep;34(9):870-7. doi: 10.1080/003655299750025327. PMID 10522604
- [Background] Aya V, Jimenez P, Munoz E, Ramirez JD. Effects of exercise and physical activity on gut microbiota composition and function in older adults: a systematic review. BMC Geriatr. 2023 Jun 12;23(1):364. doi: 10.1186/s12877-023-04066-y. PMID 37308839
- [Background] Boytar AN, Skinner TL, Wallen RE, Jenkins DG, Dekker Nitert M. The Effect of Exercise Prescription on the Human Gut Microbiota and Comparison between Clinical and Apparently Healthy Populations: A Systematic Review. Nutrients. 2023 Mar 22;15(6):1534. doi: 10.3390/nu15061534. PMID 36986264